CLINICAL TRIAL: NCT02823951
Title: Patient Real-world Clinical, Neurological, Tolerability, and Safety Outcomes for Tecfidera® and Rebif®: A Retrospective Study (PROTRACT)
Brief Title: Patient Real-world Clinical, Neurological, Tolerability, and Safety Outcomes for Tecfidera® and Rebif®
Acronym: PROTRACT
Status: Completed | Type: Observational
Sponsor: IMS HEALTH GmbH & Co. OHG (Industry)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: MS200136_0037
Record Dates: First submitted 2016-03-03; First posted 2016-07-06 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a; Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Rebif - 1 year MRI cohort: Treatment naive patients starting with Rebif, 1 year follow-up available, MRI scan available at baseline and at 12 months
  Interventions: Drug: Rebif
- Rebif - 1 year clinical cohort: Treatment naive patients starting with Rebif, 1 year follow-up available, MRI scan available at baseline
  Interventions: Drug: Rebif
- Rebif - early discontinuation cohort - tolerability: Treatment naive patients starting with Rebif, MRI scan available at baseline, discontinuation within the first treatment year due to tolerability
  Interventions: Drug: Rebif
- Rebif - early discontinuation cohort - adverse events: Treatment naive patients starting with Rebif, MRI scan available at baseline, discontinuation within the first treatment year due to adverse events
  Interventions: Drug: Rebif
- Rebif - early discontinuation cohort - disease activity: Treatment naive patients starting with Rebif, MRI scan available at baseline, discontinuation within the first treatment year due to disease activity
  Interventions: Drug: Rebif
- Tecfidera - 1 year MRI cohort: Treatment naive patients starting with Tecfidera, 1 year follow-up available, MRI scan available at baseline and at 12 months
  Interventions: Drug: Tecfidera
- Tecfidera - 1 year clinical cohort: Treatment naive patients starting with Tecfidera, 1 year follow-up available, MRI scan available at baseline
  Interventions: Drug: Tecfidera
- Tecfidera - early discontinuation cohort - tolerability: Treatment naive patients starting with Tecfidera, MRI scan available at baseline, discontinuation within the first treatment year due to tolerability
  Interventions: Drug: Tecfidera
- Tecfidera - early discontinuation cohort - adverse events: Treatment naive patients starting with Tecfidera, MRI scan available at baseline, discontinuation within the first treatment year due to adverse events
  Interventions: Drug: Tecfidera
- Tecfidera - early discontinuation cohort - disease activity: Treatment naive patients starting with Tecfidera, MRI scan available at baseline, discontinuation within the first treatment year due to disease activity
  Interventions: Drug: Tecfidera

INTERVENTIONS:
Drug: Rebif
  Groups: Rebif - 1 year MRI cohort; Rebif - 1 year clinical cohort; Rebif - early discontinuation cohort - adverse events; Rebif - early discontinuation cohort - disease activity; Rebif - early discontinuation cohort - tolerability
Drug: Tecfidera
  Groups: Tecfidera - 1 year MRI cohort; Tecfidera - 1 year clinical cohort; Tecfidera - early discontinuation cohort - adverse events; Tecfidera - early discontinuation cohort - disease activity; Tecfidera - early discontinuation cohort - tolerability

SUMMARY:
The purpose of this study is to evaluate the proportion of patients who demonstrate no medical need to discontinue therapy among DMT-naïve patients with relapsing forms of multiple sclerosis after 1 year of treatment with Rebif 44 mcg tiw or with Tecfidera 240 mg bid based on real-world data.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Clinically Isolated Syndrome (CIS) or a relapse remitting multiple sclerosis (RRMS).
2. Age between 18 - 55 years at the time of index.
3. No evidence of prior disease modifying therapy for MS.
4. Initiated treatment with either Rebif or Tecfidera at the time of index. Patient is considered to have initiated treatment if they took at least one dose. Treatment must have been initiated after the product was approved by the FDA.
5. Availability of a high quality baseline MRI brain scan, which must have occurred between 6 months prior to the index date to 2 weeks after the index date.
6. Availability of clinical data in the patient's record for the full study observation period, as defined in the primary objective.

Exclusion Criteria:

1. Pregnant at any time during the study observation period.
2. Presence of pre-existing medical conditions known to be associated with brain pathology (cerebrovascular and neurodegenerative diseases, presence of active alcohol or substance abuse).
3. Patient discontinued initial therapy prior to completing 1 year of treatment due to a reason other than disease activity, tolerability, or safety (e.g. financial, convenience, preference, etc.).
4. Phase III registrational trial patients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Treatment naive patients for Rebif or Tecfidera with at least 1 months follow-up data available from clinical chart review.
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
NEDA-2 | 12 months
  Number of patients who had no need to discontinue therapy within the first 12months after index date. Unit of measure is number of patients.
  No medical need to discontinue therapy is reached if there are no relapses and no new lesions, and no enlarging lesions and the patient did not stop the index medication due to tolerability, adverse events or disease activity. If any of the above occurs, NEDA-2 is not reached.

SECONDARY OUTCOMES:
Clinical differences between the two treatment groups | 12 months
  Comparison of number of relapses between the two treatment groups.
Neurological differences between two treatment groups | 12 months
  Comparison of number of new lesions and number of enlarging lesions between the two treatment groups. Unit of measurement is number of each lesion type.
Proportion of individuals within each treatment group who discontinued, stratified by reason | 12 months
  Proportion of individuals within each treatment group who discontinued treatment due
  * to tolerability
  * to adverse events
  * to disease activity Unit of measurement is the share of patients who discontinued compared to total patients stratified by reason of discontinuation.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - Alabama Neurology Associates, Birmingham, Alabama
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Savannah Neurology Specialists, Savannah, Georgia
  - Northshore University, Evanston, Illinois
  - OSF Multi-specialty Group d/b/a Illinois Neurological Institute, Peoria, Illinois
  - St Elizabeths/ Dragonfly Research, Brighton, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington university, St Louis, Missouri
  - University of Nebraska Medical Center, Lincoln, Nebraska
  - University of Buffalo Clinical and Translational research Center, Buffalo, New York
  - Neurological Associates of Long Island, Lake Success, New York
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Oak Clinic-Multiple Sclerosis, Uniontown, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - The university of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Blacksburg Neurology, Christiansburg, Virginia
  - MultiCare Health System, Tacoma, Washington
  - Neuroscience Group, Neenah, Wisconsin
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No